CLINICAL TRIAL: NCT01878721
Title: Positron Emission Tomography of Infection and Vasculitis (PETU)
Brief Title: Positron Emission Tomography of Infection and Vasculitis
Acronym: PETU
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Anne Roivainen, professor, Turku University Hospital
Other Study IDs: 14824
Record Dates: First submitted 2013-06-10; First posted 2013-06-17 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Infection; Vasculitis
Keywords: PET/CT; infection; vasculitis
MeSH Terms: conditions — Infections; Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Staphylococcus aureus bacteremia: PET/CT in patients with Staphylococcus aureus bacteremia
  Interventions: Radiation: PET/CT
- Salmonella spp. bacteremia: PET/CT in patients with Salmonella spp. bacteremia
  Interventions: Radiation: PET/CT
- Endocarditis: PET/CT in patients with infective endocarditis
  Interventions: Radiation: PET/CT
- Pacemaker infection: PET/CT in patients with pacemaker infection
  Interventions: Radiation: PET/CT
- Vasculitis: PET/CT in patients with vasculitis
  Interventions: Radiation: PET/CT

INTERVENTIONS:
Radiation: PET/CT — positron emission tomography/computed tomography

SUMMARY:
The purpose of this study is to evaluate the value of positron emission tomography/computed tomography in various inflammatory conditions caused by bacterial infection or vasculitis. Glucose analog FDG is sensitive to detect inflammation foci but we hypothesize that other imaging agents such as PK11195 and Ga-citrate may have added value in certain applications.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the value of PET/CT in various inflammatory conditions caused by bacterial infection or vasculitis. Our aim is to:

1. investigate whether FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET/CT and 68Ga-(Gallium-68) citrate PET/CT enable the early and accurate detection of metastatic infection foci in Staphylococcus aureus bacteremia.
2. study the usefulness of FDG PET/CT in detection of endovascular infection in bacteremia caused by Salmonella spp.
3. find an optimal FDG PET/CT protocol for detection of infectious endocarditis and metastatic infection foci related to endocarditis.
4. study the value of FDG PET/CT in the diagnosis of infection of pacemaker or implantable cardioverter defibrillator.
5. investigate the usefulness of FDG PET/CT, 68Ga-citrate PET/CT, and 11C- (carbon-11) translocator protein ligand (PK11195) PET/CT in diagnosis of vasculitis and in imaging of the magnitude of the vascular changes.

ELIGIBILITY:
Inclusion Criteria:

Adults with

* Staphylococcus aureus bacteremia or
* Salmonella spp. bacteremia or
* infective endocarditis or
* infection of pacemaker or implantable cardioverter defibrillator or
* vasculitis

Exclusion Criteria:

* underage, pregnant, breastfeeding, handicapped or prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Turku University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2011-01; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Detection of infection or vasculitis in PET images | within 1 week after starting the treatment

SECONDARY OUTCOMES:
Standardized uptake value of PET imaging agent at the site of infection or vasculitis | within 1 week after starting the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland